CLINICAL TRIAL: NCT04951193
Title: Development and Evaluation of a Brief Behavioral Activation Mobile Application for Nicotine Vaping Cessation Among Adolescent Primary Care Patients
Brief Title: Goal2QuitVaping for Nicotine Vaping Cessation Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Dahne, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00108733; 1R41DA053856-01 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Depressive Symptoms; Depression; Adolescent Behavior
MeSH Terms: conditions — Depression; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal2QuitVaping (Experimental): Participants in the Goal2QuitVaping group will be asked to download the Goal2QuitVaping app to their smartphone. Goal2QuitVaping focuses on mood management as well as on quitting vaping nicotine. Participants will be asked to use Goal2QuitVaping regularly, at least once per day, for the study duration. Participants will also be asked to complete questionnaires weekly for 4 weeks.
  Interventions: Behavioral: Behavioral Activation Therapy app
- Treatment as Usual (Other): Participants in the treatment as usual group will be provided with educational material about quitting vaping nicotine and it will be suggested that they discuss any questions about mood management and about quitting vaping with their primary care provider. The educational material is from the National Cancer Institute's SmokeFree Teen website and includes information on recognizing reasons for quitting vaping, avoiding dual use of e-cigarettes and other tobacco products, setting a quit date, understanding triggers, and accessing social support.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy app — Goal2QuitVaping focuses on tracking daily activities, recording daily mood, and identifying new activities to complete that may help improve mood. Participants will be asked to complete questionnaire measures weekly for 4 weeks following study enrollment.
  Arms: Goal2QuitVaping
Behavioral: Treatment as Usual — Participants will be provided educational material about quitting vaping nicotine with the suggestion to discuss questions with their PCP. Participants will be asked to complete questionnaire measures weekly for 4 weeks following study enrollment.
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to evaluate a mobile application (app) called "Goal2QuitVaping" to help adolescents quit vaping nicotine. Goal2QuitVaping was developed by our research team to assist with quitting vaping. Participants will be randomly assigned to either download the mobile app, "Goal2QuitVaping", or not. If provided with Goal2QuitVaping, participants will be asked to use the app regularly, at least once per day, throughout the study duration. Participants will be asked to complete electronic questionnaire measures throughout the study period. Participation in this study will take about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. age 16-20
2. vaped nicotine on ≥20 days out of the last 30
3. elevated depressive symptoms, defined as a score of ≥10 on Patient Health Questionnaire-8 (PHQ-8) during preliminary screening and the Adolescent Patient Health Questionnaire-9 (PHQ-9A) at final eligibility
4. currently own an iOS or Android smartphone
5. report willingness to utilize an app for quitting vaping nicotine (response of "yes" on yes/no item)
6. have a valid e-mail address that is checked regularly or regular access to text messages (for follow-up assessments)
7. ability to read the consent form
8. has been seen (in person or remotely) by a primary care physician within the last year

Exclusion Criteria:

1. smoked cigarettes or used other tobacco products on ≥9 days out of the last 30
2. severe visual impairment
3. currently receiving treatment for vaping or tobacco use
4. current suicidal ideation, defined as a response ≥1 on item nine of the PHQ-9A or ≥2 on item 9 of the BDI-II
5. household member currently enrolled in the study
6. inability to read the consent form

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dahne, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Goal2QuitVaping | Treatment as Usual
Started | 56 | 50
Completed | 49 | 45
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal2QuitVaping | Treatment as Usual | Total
Number analyzed (Participants) | 56 | 50 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 1 | 5
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 51 | 42 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 42 | 40 | 82
  More than one race | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Depressive Symptoms
Description: Patients will self report depressive symptoms weekly for 4 weeks via the Beck Depression Inventory-II. The range of scores possible are 0 - 63, where lower scores are indicative of lower symptoms of depression. This outcome will measure change from baseline at week 4.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal2QuitVaping | Treatment as Usual
Number analyzed (Participants) | 50 | 49
score on a scale | -9.50 (9.54) | -8.30 (9.72)

2. Primary Outcome: Average Vapes Per Day at Week 4
Description: Assessed using the Timeline Followback during each weekly assessment. Average vapes per day at week 4.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: vapes per day
Arm/Group | Goal2QuitVaping | Treatment as Usual
Number analyzed (Participants) | 50 | 49
vapes per day | 9.42 (16.11) | 10.17 (11.89)

3. Primary Outcome: E-cigarette Dependence
Description: Assessed at baseline via the 10-item Penn State Electronic Cigarette Dependence Index (ECDI). Change from baseline at week 4. The scores range from 0-20 with 0-3= not dependent, 4-8 low dependence, 9-12 medium dependence, 13+ = high dependence.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal2QuitVaping | Treatment as Usual
Number analyzed (Participants) | 50 | 49
score on a scale | -2.19 (3.30) | -2.38 (2.86)

4. Primary Outcome: Number/Duration of Quit Attempts
Description: Assessed during the Timeline Followback. Total number of quit attempts across all 4 weeks
Time Frame: Across all 4 weeks
Measure: Mean (Standard Deviation); unit: number of quit attempts
Arm/Group | Goal2QuitVaping | Treatment as Usual
Number analyzed (Participants) | 50 | 49
number of quit attempts | 5.00 (4.35) | 4.00 (4.11)

5. Primary Outcome: 7-day Point Prevalence Abstinence
Description: Assessed during the Timeline Followback. At any point during the study across all 4 weeks.
Time Frame: At any point during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Goal2QuitVaping | Treatment as Usual
Number analyzed (Participants) | 50 | 49
Participants | 14 | 15

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Goal2QuitVaping | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/50
Other Adverse Events (participants affected / at risk) | 0/56 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04951193/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04951193/ICF_000.pdf